CLINICAL TRIAL: NCT07373925
Title: Effect of Kinesio Taping Versus Dry Cupping Therapy in Treatment of Thoracic Kyphosis: A Randomized Control Trial
Brief Title: Kinesio Taping Versus Dry Cupping Therapy in Treatment of Thoracic Kyphosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Alaa Eldeen Sultan, Principal investigator: Aya Alaa Eldeen Sultan, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T/REC/012/006192
Record Dates: First submitted 2026-01-21; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Thoracic Kyphosis
Keywords: Kinesio taping; Dry Cupping Therapy; Thoracic Kyphosis

STUDY DESIGN:
Intervention Model Description: Kinesio taping and Dry Cupping Therapy
Who Masked: Outcomes Assessor
Masking Description: sealed envelopes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio taping (Experimental): 16 participants will receive Kinesio taping once a week for 4 weeks + traditional treatment
  Interventions: Other: Kinesio taping; Other: Conventional treatment
- Dry Cupping Therapy (Experimental): 16 participants will receive Dry Cupping Therapy 3 times a week for 4 weeks + traditional treatment
  Interventions: Other: Dry Cupping Therapy; Other: Conventional treatment
- Conventional treatment (Active Comparator): 16 participants will receive traditional treatment
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Kinesio taping — The subjects in this group will be treated with KT in addition to the traditional treatment for thoracic kyphosis. Elastic tape (Kinesio tape, Kinesio® Tex Classic, Kinesio Holding Corporation, New Mexico, USA) 5 cm in width will be applied on the upper back of participants by a certified physiotherapist. When applying the tape, the participants will be in an upright standing position with both arms along the side of the body in a relaxed position. Taping will be applied from a starting point at the anterior aspect of the acromioclavicular joint and will be applied across the spinous process at T6 with the tape ending around T12 paraspinal muscle. The elastic tape will be applied with a stretch of approximately 150 %, .Taping will not be taken off for four days. After day four, it will be taken off and the skin will be rested for two days. Taping application will be repeated on day 7. The patients in this group will be followed for four weeks.
  Arms: Kinesio taping
Other: Dry Cupping Therapy — Participants in this group will receive three sessions per week for four weeks. Two sessions will include cupping therapy in addition to conventional treatment, while one session will consist of conventional treatment only. Six stationary cups will be placed directly around the thoracic spine three cups on each side of the spine. Reusable acrylic cups of medium diameter (3.5 cm) will be used for each individual at each session. The participant will be asked to lie prone. Before beginning the session, if any signs of dehydration are identified by the therapist, coconut oil will be applied to the region in order to hydrate the skin. cups will initially be applied through two suctions by the hand pump, "moderate" suction, which generates a negative pressure of approximately 300 millibar. For participants who report considerable discomfort, the pressure will slightly be minimized according to the individual sensation. cups will be positioned around the thoracic region for 10 Min.
  Arms: Dry Cupping Therapy
Other: Conventional treatment — The participants in this group will receive conventional treatment that will include advices, stretching, strengthening and functional exercises 3 sessions a week for 4 weeks.

SUMMARY:
This study will be conducted to investigate the effect of Kinesio taping versus dry cupping therapy in the treatment of thoracic kyphosis

DETAILED DESCRIPTION:
Kyphosis is defined as an increase in the forward curvature of the spine that is seen along the sagittal plane. When the forward curvature becomes excessive, this is called hyperkyphosis. The curvature can be a normal variance when presented in the thoracic spine or in excess be a cause for instability and concern. The natural history of kyphosis is not exactly well known. Kinesio Taping (KT) stands out as one such modality proposed to manage musculoskeletal disorders (MSK) disorders. First developed in the 1970s by Dr. Kenzo Kase, It is touted for pain relief, increased range of motion (ROM), and muscle relaxation. As such, it is widely used, not only among athletes but also in clinical medicine Another traditional technique is known as dry cupping therapy that involve the application of cups to create localised negative pressure on the skin, has been utilised for over four thousand years. Its use spans various conditions, including musculoskeletal pain. Dry Cupping has traditionally carried folkloric, cultural, religious, and spiritual significance within various societies It is used for health promotion, prophylaxis and treatment of a variety of diseases around the world. It is a well-recognized traditional method for managing medical conditions. Currently, the scope of cupping therapy is expanding, and a growing body of research is providing additional evidence-based data for the further advancement of this therapy in the treatment of a variety of diseases. It has gained popularity and acceptance as a method of treating pain as well as sports injuries and other medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with thoracic kyphosis angle > 40° diagnosed by a medical doctor will be selected from Damietta University's clinic of physical education faculty.
* Subjects from both genders with an age range between 18 and 30 years .
* Subjects who are physically active in physical education sessions

Exclusion Criteria:

* Subjects with medical conditions that restrict activity.
* Those who received exercise intervention for kyphosis.
* Structural thoracic kyphosis, defined as thoracic kyphosis that did not partially or completely disappear during prone extension, as assessed by a physical therapist.
* Medical history of spinal fracture, spinal surgery, shoulder joint injury or pelvic injury.
* Other spinal diseases; presence of scoliosis on Adam's forward bend test.
* Spinal kyphosis due to visible thoracic deformity.
* Subjects undergoing professional sports training.
* Skin disease (dermatitis, psoriasis), neurological disease or cancer.
* Using anticoagulants or nonsteroidal antidepressants.
* Inflammatory or rheumatologic disorders of the spine.
* Severe cardiopulmonary disease, rheumatic disease or pregnancy.
* Have a pacemaker or metal implants.
* Do not understand the written consent form.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Level | up to 4 weeks
  A visual analogue scale (VAS) will be used to measure the intensity of pain. With a score of 0 for no pain and 10 for the worst pain ever, this psychometric response scale, which measures pain intensity based on numerical values, is 10 cm or 100 mm in length. The interclass correlation ranges for the VAS, a validated and dependable measure of pain intensity, are 0.95 to 0.98. Patients rated their level of pain as mild if they scored 3.4 or less, moderate if they scored 3.5 to 7.4, and severe if they scored 7.5 or higher.

SECONDARY OUTCOMES:
Thoracic-curve angle | up to 4 weeks
  The digital inclinometer will be used to measure thoracic-curve angle. It is a precision instrument designed to measure angles of slope, tilt, or inclination. The digital inclinometer is becoming a popular tool to assess the musculoskeletal system, including the antero-posterior curvatures of the spine, in both clinical practice and research. The digital inclinometer is a valid and reliable instrument for measuring thoracic kyphosis and can be used for regular screening.